CLINICAL TRIAL: NCT05642013
Title: SHort Interval Full Two-stage Implant Exchange
Acronym: SHIFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL22_0231
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Prosthetic-joint Infection
Keywords: prosthetic joint infection; knee; hip; two-stage exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospective group (Experimental): 50 patients prospectively included with early prosthesis reimplantation
  Interventions: Procedure: Early prosthesis reimplantation
- Retrospective group (Other): Last 50 patients with hip or knee prosthetic-joint infection managed with classical two-stage implant exchange
  Interventions: Other: Retrospective analysis of medical records

INTERVENTIONS:
Procedure: Early prosthesis reimplantation — Early prosthesis reimplantation, within 16 to 30 days after implants removal
  Arms: Prospective group
Other: Retrospective analysis of medical records — Analysis of 50 records of operated patients managed with classical two-stage implant exchange
  Arms: Retrospective group

SUMMARY:
This study is a prospective bicentric feasibility study, which aims to evaluate the feasibility of a two-stage full implant exchange with early prosthesis reimplantation between 16 and 30 days after implants removal for hip or knee prosthetic joint infection.

This study concern 50 patients, prospectively included and compared to the last 50 patients with hip or knee PJI managed with classical two-stage implant exchange.

The duration of the study is 42 months.

DETAILED DESCRIPTION:
Prosthetic joint infection (PJI) is a rare but severe complication, with long and complex medico-surgical procedures ang high morbidity. Two-stage full implant exchange is commonly used for PJI, but the best time for prosthesis reimplantation remains unclear. Late reimplantation leads to prolonged immobilization, which can cause decubitus complications and altered joint functionnality.

The hypothesis is that reimplantation between 16 and 30 days after implants removal, earlier than suggested by some relatively old recommandations, associated with 12 weeks antibiotic therapy is a safe and efficient option, allowing shorter immobilization susceptible to improve joint functionnality.

The principal aim of this study is to evaluate the feasibility of a two-stage full implant exchange with early prosthesis reimplantation.

50 patients with knee or hip PJI eligible for two-stage implant exchange will be prospectively included in two french centers.

Surgical procedure will be standardized, with prothesis reimplantation within 16 to 30 days after implants removal, associated with 12 weeks adaptated antibiotherapy according to french recommendations.

Patients will be compared to the last 50 patients with hip or knee PJI managed with classical two-stage implant exchange in these centers until december 2021 (retrospective group).

Follow up consists of 7 clinical evaluations, from inclusion until month15 after prosthesis removal.

ELIGIBILITY:
Inclusion Criteria:

Prospective group:

* Patient over 18 years old
* Patient managed for a definite osteoarticular infection in a hip or knee prosthesis according to EBJIS definitions (2021) Clinical definition : fistula communicating with the prosthesis, prosthesis exposed / Or biological ≥ 2 samples positive for the same microorganism / And/ or 3000 leukocytes or > 80% of PNN on the synovial fluid / Or histological: visible microorganism, > or = 5 PNN on 5 HPN
* Patient with an indication for 2-stage surgery:

A Impossibility of conservative treatment : infection occurring more than 4 weeks after prosthesis implantation, fistula, documented resistant germ, loosened prosthesis / B Unsuitable 1-stage change: recurrence after 1-stage management, precarious bone capital, documented resistant microorganism, infection without prior microbiological documentation, fistula, surgeon's assessment in disfavor

- Effective contraception during the research period for fertile women of childbearing age

Retrospective group :

* Patient managed before 31/12/2021 for a definite osteoarticular infection in a hip or knee prosthesis according to EBJIS definitions (2021) Clinical definition : fistula communicating with the prosthesis, prosthesis exposed Or biological ≥ 2 samples positive for the same microorganism And/ or 3000 leukocytes or > 80% of PNN on the synovial fluid Or histological: visible microorganism, > or = 5 PNN on 5 HPN
* Patient managed by 2 "long" stage surgery with reimplantation time > 6 weeks with an evolutionary follow-up of at least 15 months after the end of antibiotics

Exclusion Criteria:

Prospective group :

* Indication for conservative treatment, 1-stage or 2 long stage surgery
* Reimplantation by another surgical approach requiring complete skin closure of the initial scar
* Other surgeries scheduled within 30 days of removal
* Participation in another interventional treatment study and/or in an exclusion period due to participation in another protocol
* Subject not affiliated with a social security plan or beneficiary of such a plan
* Failure to obtain written informed consent
* Patient with a legal protection measure (guardianship, curatorship)
* Patient under justice safeguard
* Pregnant or breastfeeding woman

Retrospective group :

- Refusal to participate

Study exit criteria

* Bacteriological samples positive for fungi
* Infection not retained after analysis of samples (no sufficient clinical or biological criteria according to EBJIS definition)
* Withdrawal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2026-04-23 (Estimated); Study Completion 2027-07-23 (Estimated)

PRIMARY OUTCOMES:
Rate of eligible patients included and benefiting from the standardized protocol without major deviations | At 3 months follow-up
  Number of eligible patients having been included in the study having benefited from the standardized protocol without major deviations / number of eligible patients according to surgeons or doctors during consultations and hospitalization in orthopedic or infectious disease departments

SECONDARY OUTCOMES:
Rate of eligible patients included | At 3 months follow-up
  Number of eligible patients included in the study / number of eligible patients according to surgeons or doctors during consultations and hospitalization in orthopedic or infectious disease departments
Rate of clinical cure | At 15 months follow-up
  Number of patients included without signs of infectious relapse to the same germ or persistence of the initial infection at M15 / number of patients included who benefited from the standardized protocol without major deviations., compared to clinical cure rate in retrospective group
Rate of re-infection with a different microorganism (superinfection) during follow-up and up to M15 | At 15 months follow-up
  Number of patients who presented a reinfection according to the EBJIS criteria with a germ different from the initial organism(s) during follow-up / number of patients included who benefited from the standardized protocol without major deviations, compared to reinfection rate in retrospective group
Length of stay | At 15 months follow-up
  Cumulative length of stay in hospital (medicine or surgery wards) or in follow-up care compared to cumulative length of stay in retrospective group
Articular functionnality | At 6 months follow-up
  Knee Society Score or Harris Hip Score
Articular functionnality | At 15 months follow-up
  Knee Society Score or Harris Hip Score
Quality of life auto-evaluation score | At inclusion
  EQ-5D-5L score (auto-questionnary)
Quality of life auto-evaluation score | At 3 months follow-up
  EQ-5D-5L score (auto-questionnary)
Quality of life auto-evaluation score | At 15 months follow-up
  EQ-5D-5L score (auto-questionnary)
Antibiotics tolerance | From inclusion to 3 months follow-up
  Evaluation of antibiotics tolerance by clinical +/- biological evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie PANSU, MD, Principal Investigator — Infectious Diseases department, Montpellier university hospital
Locations (2):
- France (2):
  - CHU de Montpellier - Hôpital Saint-Eloi, Montpellier
  - CH de Sète - Hôpitaux du bassin de Thau, Sète

IPD SHARING:
Plan to Share IPD: No